CLINICAL TRIAL: NCT07162220
Title: The Effect of a Mobile Game Application Developed for Children With Chronic Renal Failure on Disease Management
Brief Title: The Effect of a Mobile Game Application on Children With CRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Sakarya Applied Sciences University (Other); Tarsus University (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, Banu Terzi, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: CRF_2022/04
Record Dates: First submitted 2025-08-23; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Child, Only; Chronic Renal Failure in Children; Gambling; Disease; Management
Keywords: chronic renal failure; child; mobile game; disease management
MeSH Terms: conditions — Gambling; Disease; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant
Masking Description: To control statistical bias, the data were transferred to a computer by an independent researcher, coded as groups A and B, and entered into the database. After the data were analyzed by a statistician and a statistical report was written, the control and research groups were reported by the coder.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine application (Other): No procedures outside of the clinic's routine were performed on the children in the control group. As part of the clinic's routine education program, information about kidney function, CKD, nutrition, exercise, medications, and stress management is provided verbally by a nephrology clinic nurse in approximately 20 minutes. The Chronic Kidney Disease Information Form, the Healthy Lifestyle Belief Scale for Adolescents, and the Child's Attitude Toward Their Own Illness Scale were administered to the children before the education program, after the program, and at the end of the first and third months, and the relevant clinical parameters were measured.
  Interventions: Other: The clinic's routine education program
- Intervention (Experimental): A mobile game application was downloaded onto the phones of the children participating in the study group. Before starting the mobile game, after completing the application, and at the end of the first and third months, the Chronic Kidney Disease Information Form, the Healthy Lifestyle Belief Scale for Adolescents, and the Child's Attitude Toward Their Own Illness Scale were administered, and relevant clinical parameters were measured. At the end of the study, the Mobile Application Usability Scale was also administered.
  Interventions: Device: Mobile game app

INTERVENTIONS:
Other: The clinic's routine education program — As part of the clinic's routine education program, information about kidney function, CKD, nutrition, exercise, medications, and stress management is provided verbally by a nephrology clinic nurse in approximately 20 minutes.
  Arms: Routine application
Device: Mobile game app — The mobile game software developed for patients with chronic renal failure contains information for children on daily life activities such as nutrition, exercise, personal hygiene, etc.
  Arms: Intervention

SUMMARY:
The aim of this study was to investigate the effect of a mobile game application developed for children with Chronic Renal Failure (CRF) on disease management.

The study was a randomized controlled trial. The study sample consisted of 68 children diagnosed with CRF, including the Mobile application (n:34) and Control group (n:34). In the study, a mobile game was developed for children diagnosed with CRF aged 11-14 years. Data Collection Form, Clinical Parameters Follow-up Form, Information Form on Chronic Renal Failure, Healthy Lifestyle Belief Scale for Adolescents, Child's Attitude Toward His/her Disease Scale and Mobile Application Usability Scale were used to collect the data.

ELIGIBILITY:
Inclusion Criteria:

* (a) 11-14 years old
* (b) Being monitored with a diagnosis of Chronic Kidney Failure
* (c) having the ability to read, write, and understand Turkish
* (d) having a phone/tablet with mobile game download capability
* (e) volunteering to participate in the study
* (f) being willing to participate in the study.

Exclusion Criteria:

* (a) having mental, neurological, or communication problems
* (b) being on hemodialysis
* (c) communication, mental or neurological problems
* (d) being on peritoneal dialysis
* (e) having previously attended planned training on CRF

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
BMI | 3 months
  BMI in kg/m^2
Blood pressure | 3 months
Pulse rate | 3 months
Level of knowledge regarding chronic renal failure | 3 months
  The information form consists of 25 questions. The information form has been created with two answers, correct and incorrect. Correct answers are worth 1 point, while incorrect answers are worth 0 points, and the form is evaluated based on the total score. A reliability analysis was performed using Kuder Richardson 20 (KR-20) to evaluate whether the items that make up the question form form a whole.
Healthy Lifestyle Belief Level for Adolescents | 3 months
  The scale emphasizes beliefs related to various aspects of maintaining a healthy lifestyle. The scale has a total of 16 items. The scale has three subscales: health beliefs, physical activity, and nutrition. The health beliefs subscale is composed of items 4, 5, 6, 11, 12, 13, and 16; the physical activity subscale includes items 2, 7, 9, 14, and 15; and the nutrition subscale comprises items 1, 3, 8, and 10. The scale, prepared according to the five-point Likert system, is answered on a scale of "1=Strongly Disagree, 5=Strongly Agree." A minimum of 16 and a maximum of 80 points can be obtained from the entire scale. An increase in the score obtained from the scale indicates an increase in adolescents' belief in healthy living.
Child's Attitude Towards Their Own Illness | 3 months
  The Child's Attitude Toward Their Own Illness Scale is a 13-item measure developed to assess children's feelings and thoughts about having a chronic illness. Participants respond to the scale items using a 5-point Likert scale: "never, not often, sometimes, often, and very often." Items 1, 2, 3, 4, 5, 7, 9, 11, and 13 are reverse-coded. When evaluating the scale, the scores obtained from the 13 items are summed and divided by the number of items. The total score range is min: 1 to max: 5. Scores of 1 and 2 indicate a negative attitude, 3 indicates a neutral attitude, and 4 and 5 indicate a positive attitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No